CLINICAL TRIAL: NCT06197711
Title: The Short-term Effects of PRISMA on Mental Health
Acronym: PRISMA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: ETH Zurich (Other); The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC-Nr. 2023-01378
Record Dates: First submitted 2023-12-04; First posted 2024-01-09 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Psychological Distress; Anxiety; Depression; Suicidal Ideation
Keywords: PRISMA; psychological intervention; psychological distress; inmates; pretrial detention
MeSH Terms: conditions — Anxiety Disorders; Depression; Suicidal Ideation | interventions — mesoglycan

STUDY DESIGN:
Intervention Model Description: The RCT will inform about the effect of PRISMA. Of the projected 5'100 people entering pretrial detention during the enrollment window, it is expected that roughly 43% (or 2'194 individuals) will be eligible for PRISMA and roughly 65% (or 3'316 individuals) will be eligible for the proactive social services intervention, respectively. Thus, it is expected that 1'428 individuals to be eligible for both interventions and, hence, constitute randomization sample C. This means that 766 individuals will be eligible for PRISMA only and 1'888 individuals for proactive social services only. 1'018 individuals will not be eligible for any of the two interventions.
  For the analysis, observations from the REGULAR PRETRIAL and the PRISMA group from randomization samples A and C, respectively, will pooled. This leaves N = 1480 participants who will be involved in the RCT (assigned to either receiving the PRISMA intervention (N=740) or control condition (N = 740)).
Who Masked: Outcomes Assessor
Masking Description: All instruments and questions will be administered online.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention, PRISMA, addresses the issue of poor mental health of inmates during pretrial detention and after release. PRISMA has been adapted for the context of the model trial from Problem Management Plus (PM+). PRISMA has a total of four sessions provided during the first two weeks after entry such that most inmates can benefit from it before their potential release. The four sessions involve stress management, problem solving, meaningful activities (behavioral activation, and strengthening social support) and relapse prevention (staying well, looking forward). Additionally, participants will receive 2 booster sessions, 4 and 9 weeks after the final session, when most inmates will already have been released from jail.
  Interventions: Behavioral: PRISMA
- Control group (No Intervention): REGULAR PRETRIAL: participants in this group experience the same pretrial system, conditions, and services that they would have experienced if the RCT did not exist. They will not be offered PRISMA or extended social services, but they can still access social services upon request as well as medical support through the jails' health services.

INTERVENTIONS:
Behavioral: PRISMA — PRISMA has been developed adapting PM+, a brief, psychological intervention program based on CBT techniques that are empirically supported and formally recommended by the WHO. The adapted manual was developed to tailor the sessions to the structure of the Swiss prison system and the needs of inmates of jails in Switzerland. PRISMA involves the following elements: stress management, problem-solving, meaningful activities and relapse prevention
  PRISMA has four core features:
  * Evidence-based problem-solving strategies
  * Brief and easy to learn
  * Delivered by lay-helpers ("trainers")
  * Transdiagnostic, addressing depression, anxiety, stress, and practical problems as defined by participants; PRISMA has four sessions.
  Arms: Intervention group

SUMMARY:
Given the high prevalence of mental health issues, such as anxiety and depression, in pretrial detainees, the Swiss Federal Justice Department (SFJD) approved a model trial ("Modellversuch Untersuchungshaft", MV). The MV will be carried out in 11 pretrial detention facilities in the cantons of Zurich and Bern and aims to improve the wellbeing and social integration of individuals in pretrial detention. As part of the MV the investigators are evaluating the impact of two interventions using a randomized controlled trial (RCT). The first intervention, "Prison Stress Management" (PRISMA), addresses the issue of poor mental health of inmates during pretrial detention and after release. PRISMA is a scalable World Health Organization (WHO)-developed psychological intervention based on cognitive-behavioral therapy (CBT) program and goes beyond the status-quo mental health support offered in jails. Currently, only inmates with severe mental health problems are referred to the psychiatric ward of the health services provided in jails and no continuation of support is offered after the transition to the outside world. The second intervention (SOCIAL) uses extended social services to address potential disruptions incarceration might cause in detainees' social and economic lives. The isolation from the outside world implies that detainees might lose their jobs and housing, their relationships with their family and friends are strained, all factor hindering re-integration into society and taxing their mental wellbeing. This project will provide much needed insights to criminal justice authorities to design detention facilities and the detention experience in ways that empower incarcerated individuals to cope with the disruptions and psychological stress that come along with their detention.

DETAILED DESCRIPTION:
The RCT will inform about the effect of PRISMA.

The sample size is determined by the enrollment window (from November 27, 2023 to September 30, 2026). Based on historical data, the investigators expect roughly 5,100 subjects to enter pretrial detention in the cantons of Zurich and Bern during this period.

Of the projected 5'100 people entering pretrial detention during the enrollment window, it is expected that roughly 43% (or 2'194 individuals) will be eligible for PRISMA and roughly 65% (or 3'316 individuals) will be eligible for the proactive social services intervention, respectively. Thus, it is expected that 1'428 individuals (or 28% = 43% of 65%) to be eligible for both interventions and, hence, constitute randomization sample C. This means that 766 individuals (= 2'194 - 1'428) will be eligible for PRISMA only (randomization sample A) and 1'888 individuals (= 3'316 - 1'428) for proactive social services only (randomization sample B). 1'018 (= 5'100 - 1'428 - 766 - 1'888) individuals will not be eligible for any of the two interventions. If samples are split with equal probability into experimental groups, the investigators expect the following group sizes:

Randomization sample A:

REGULAR PRETRIAL: 383 PRISMA: 383

Randomization sample B:

REGULAR PRETRIAL: 944 SOCIAL: 944

Randomization sample C:

REGULAR PRETRIAL: 357 PRISMA: 357 SOCIAL: 357 PRISMA & SOCIAL: 357 For the analysis, observations from the REGULAR PRETRIAL and the PRISMA group from randomization samples A and C, respectively, will be pooled. This leaves N = 1480 participants who will be involved in the RCT (assigned to either receiving the PRISMA intervention (N=740) or control condition (REGULAR PRETRIAL) (N = 740)).

This preregistration focuses on the short-term effects of PRISMA on mental wellbeing and therefore only considers the REGULAR PRETRIAL and PRISMA treatment arms. See "Mental Health Intervention and Social Service in Pretrial Detention" on www.socialscienceregistry.org for preregistration of the other treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* • Entering pretrial detention inmate in any of the 11 pretrial detention facilities in the Cantons of Zurich and Bern

  * aged ≥ 18 years

Exclusion Criteria:

* Not fluently speaking any of the nine languages in which PRISMA is offered: German, Albanian, Arabic, English, French, Italian, Romanian, Serbian/ Croatian, Spanish

  * Acute suicidality
  * Not interested in PRISMA and its randomized evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1480 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in psychological distress | Three weeks (primary outcome) after intake; 10 weeks after the intervention
  The primary outcome is mental health at three weeks as measured by the combined two scales. Subscales can be calculated for depression measured by Patient Health Questionnaire - 9 (PHQ9) and anxiety, measured by Generalized Anxiety Disorder-7 (GAD-7). A higher score on the PHQ9 (range = 1 - 27) means a greater severity of depressive symptoms. A higher score on the GAD-7 (range = 0 - 21) means a greater severity of anxiety symptoms.

SECONDARY OUTCOMES:
Suicidal ideation | Screening, 3 weeks follow-up assessment, 10 weeks after the intervention
  Suicidal Ideation is measured using an adapted version of the Suicidal Ideation Attribution Scale (SIDAS), a brief measure of severity of suicidal ideation assessing frequency, controllability, closeness to attempt, level of distress associated with the thoughts and impact on daily functioning. It consists of 3 items rated on an 11-point scale (0 = "Never" to 10 = "Always").
Assessing the extent to which the strategies taught in PRISMA are used before and after the study participation with the Reducing Tension Checklist | 3 weeks follow-up assessment (after intake)
  The outcome is measured with a six-item scale that was developed to assess the extent to which the participants perceive that they use the specific strategies, which are trained during the study intervention. The items are rated on a scale from 0 to 4. Higher scores represent greater usage of the strategies.
General Health | 3 weeks after intake, 10 weeks after the intervention
  Assessment of the general health as assessed with Patient Reported Outcomes Measurement and Information System (PROMIS) with two global physical health items (GPH-2 (Hays et al., 2017). The two items are rated on a 5-point Likert scale from 1 to 5 (range 2-10). Higher scores represent better global health.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] van Spijker BA, Batterham PJ, Calear AL, Farrer L, Christensen H, Reynolds J, Kerkhof AJ. The suicidal ideation attributes scale (SIDAS): Community-based validation study of a new scale for the measurement of suicidal ideation. Suicide Life Threat Behav. 2014 Aug;44(4):408-19. doi: 10.1111/sltb.12084. Epub 2014 Feb 24. PMID 24612048